CLINICAL TRIAL: NCT04935632
Title: Perioperative Collection of Temperatures and Hypothermia (Recueil périOpératoire Des Températures et de l'Hypothermie - ROTHY)
Brief Title: Perioperative Collection of Temperatures and Hypothermia
Acronym: ROTHY
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ROTHY
Record Dates: First submitted 2021-06-11; First posted 2021-06-23 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Hypothermia; Hypothermia; Anesthesia; Hypothermia, Accidental
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Before implementation: Prior to the implementation of the measures resulting from the SFAR recommendations on the prevention of accidental perioperative hypothermia
- After implementation: After implementation of the measures resulting from the SFAR recommendations on the prevention of accidental perioperative hypothermia
  Interventions: Behavioral: prevention training
- at a distance from the implementation: Approximately 8 months after implementation of the measures resulting from the SFAR recommendations on the prevention of accidental perioperative hypothermia.
  Interventions: Behavioral: prevention training

INTERVENTIONS:
Behavioral: prevention training — Evaluate the impact of hypothermia prevention training on the proportion of patients hypothermic patients in the operating room
  Groups: After implementation; at a distance from the implementation

SUMMARY:
Accidental perioperative hypothermia is a frequent complication of anesthesia that favors the occurrence of infections, bleeding and perioperative cardiovascular accidents, and is responsible for perioperative excess mortality. Although preventive measures are widely used, it remains very frequent in France. This observation led a group of experts to draft, under the aegis of the Société Française d'Anesthésie et de Réanimation (SFAR), several recommendations aimed at improving the prevention of perioperative accidental hypothermia.

Perioperative hypothermia is defined as a core body temperature below 36.0 ° Celsius.

This study aims to evaluate the impact of hypothermia prevention training on the proportion of hypothermic patients in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* surgeries performed at the Centre Léon Bérard

Exclusion Criteria:

* Digestive endoscopy, interventional radiology, brachytherapy (operating rooms outside the central operating room)
* Patient who decline to participate in the study
* Active systemic infection
* Hyperthermic Intraperitoneal Chemotherapy (HIPEC) or Intrathoracic Chemotherapy (HITeC)
* Deprivation of liberty
* operation performed under local anesthesia only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated on at the Léon Bérard Centre, whether for scheduled, emergency or outpatient surgery
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypothermia | Up to 24 hours
  From the time of entry into the operating room to the time of exit from the operating room. Hypothermia is defined as a core body temperature below 36°Celsius (presence or absence).

SECONDARY OUTCOMES:
Incidence of hypothermia in the post-anesthesia care unit (PACU) | Up to 24 hours
  From the time of entry into the PACU, hypothermia is defined as a core body temperature below 36°Celsius (presence or absence).
Tympanic temperature in the post-anaesthesia care unit (PACU) | Up to 24 hours
  From the time of entry into the PACU to the time of exit from the PACU.
Intraoperative tympanic temperature | Up to 24 hours
  From the time of entry into the operating room to the time of exit from the operating room.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sari S, Aksoy SM, But A. The incidence of inadvertent perioperative hypothermia in patients undergoing general anesthesia and an examination of risk factors. Int J Clin Pract. 2021 Jun;75(6):e14103. doi: 10.1111/ijcp.14103. Epub 2021 Feb 28. PMID 33616248